CLINICAL TRIAL: NCT05616507
Title: A Phase II Trial of Oligo-Fucoidan in Radiation Induced Ling Injury
Brief Title: Oligo-Fucoidan Decrease Lung Radiation Damage
Acronym: FIRILI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB109-196-A
Record Dates: First submitted 2022-04-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-04

CONDITIONS: Radiation Toxicity
Keywords: radiation pneumonitis; fucoidan; radiation induced cardiac toxicity
MeSH Terms: conditions — Radiation Injuries; Radiation Pneumonitis | interventions — fucoidan

STUDY DESIGN:
Intervention Model Description: Study Type : Interventional (Clinical Trial) Actual Enrollment : 100 participants Allocation: Randomized Intervention Model: Parallel Assignment, matching sex, age, and performance status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): It is recommended to consume on an empty stomach, 2 servings per day, a total of 8 tablets, which can be eaten at one time or in divided doses. If it is difficult to swallow, the powder in the capsule can also be taken out and mixed with food or liquid food.
  Interventions: Dietary Supplement: fucoidan
- Arm B (No Intervention): observation

INTERVENTIONS:
Dietary Supplement: fucoidan — It is recommended to consume on an empty stomach, 2 servings per day, a total of 8 tablets, which can be eaten at one time or in divided doses. If it is difficult to swallow, the powder in the capsule can also be taken out and mixed with food or liquid food.
  Arms: Arm A

SUMMARY:
Fucoidan is FDA approved and in common use for treatment of angina. These studies will advance that work to human use. Successful mitigation of lung radiation damage and heart toxicity will improve the quality of life in veterans and non-veterans who are treated for lung cancer by radiation, and may also improve cure rates of radiation therapy for lung cancer.

DETAILED DESCRIPTION:
This project will test the effect of Fucoidan to mitigate the lung damage that can occur as a side effect of radiation therapy for lung cancer. Thousands of veterans develop lung cancer every year, and are treated by radiation therapy. Studies of lung radiation injury in laboratory animals show that with Fucoidan, investigators can significantly reduce the severity of lung fibrosis and heart toxicity.1,2 Fucoidan is FDA approved and in common use for treatment of angina. These studies will advance that work to human use. Successful mitigation of lung radiation damage and heart toxicity will improve the quality of life in veterans and non-veterans who are treated for lung cancer by radiation, and may also improve cure rates of radiation therapy for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ages Eligible for Study: 20-90 years old
2. Men and women undergoing radiation therapy for lung cancer，no matter the radiation therapy is for curing or for palliating.
3. Karnofsky performance status，KPS > 70
4. Absolute Neutrophils > 1000/mm^3
5. Platelets > 75,000/mm^3
6. Hematocrit > 25%.
7. Liver and kidney function tests will be within normal range
8. Baseline blood pressure will be systolic > 110 mmHg sitting

Exclusion Criteria:

1. Patients who get lung cancer but no need or without the willingness of radiation therapy
2. Patients who are taking antiHTN drugs
3. Women of pregnant, lactating, childbearing potential, or with the intention of becoming pregnant
4. Patients who are presently participating in another clinical study (except for follow-up surveys for study outcomes)
5. Patients who are judged to be ineligible for study entry by the investigator or subinvestigator

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 20-90
Enrollment: 100 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Radiation Pneumonitis | 6 months
  The clinical occurrence and grade of radiation pneumonitis, by National Cancer Institute Common Terminology Criteria Adverse Event grading ( NCI CTCAE) (Grade 0-5)

SECONDARY OUTCOMES:
Number of Participants With Radiation Pneumonitis | one year
  The clinical occurrence and grade of radiation pneumonitis, by National Cancer Institute Common Terminology Criteria Adverse Event grading ( NCI CTCAE) (Grade 0-5)
Number of Participants With Radiation Pneumonitis | two year
  The clinical occurrence and grade of radiation pneumonitis, by National Cancer Institute Common Terminology Criteria Adverse Event grading ( NCI CTCAE)(Grade 0-5)

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Yuan Wu, Study Director — Asia University, Taiwan
Locations (1):
- Szu-Yuan Wu, Taipei, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
study completed
Supporting Information: Study Protocol
Time Frame: data will become available on April 30 2022.
Access Criteria: requirement with official application